CLINICAL TRIAL: NCT03838185
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Single Ascending Oral Doses of J147 in Healthy Young Volunteers and Healthy Elderly Volunteers
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics of Single Ascending Oral Doses of J147
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abrexa Pharmaceuticals, Inc. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABRJ147001
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer's Disease
Keywords: Dementia; Neurodegenerative Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases | interventions — J147

STUDY DESIGN:
Intervention Model Description: Subjects will receive a single dose of J147 or placebo in a fasted state. The dose levels are planned to be administered in ascending order. Progression to the next dose level, and dose selection, will be based on all available safety and tolerability data up to at least 48 hours post-dose and available PK data (up to at least 24 hours post-dose) from a minimum of 6 subjects (J147 n ≥4) in the preceding dose cohort. Healthy elderly subjects will receive doses that have been found to be safe in healthy young subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Drug (Experimental): Healthy young male subjects will receive a single ascending oral dose of J147 following an overnight fast of at least 8 hours. Healthy elderly subjects will receive doses that have been found to be safe in healthy young subjects.
  Interventions: Drug: J147
- Placebo (Placebo Comparator): Subjects will receive a single oral dose of placebo with 240 mL non-carbonated water in the morning following an overnight fast of at least 8 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: J147 — Single oral dose of J147
  Arms: Study Drug
Drug: Placebo — Single oral dose of corn oil
  Arms: Placebo

SUMMARY:
This Phase I clinical study is a randomized, double-blind, placebo-controlled, parallel-design study to thoroughly assess the safety profile and PK properties of J147 in healthy subjects. The study will include single ascending dose (SAD) in healthy young and elderly subjects.

DETAILED DESCRIPTION:
This Phase I clinical study is a randomized, double-blind, placebo-controlled, parallel-design study to thoroughly assess the safety profile and PK properties of J147 in healthy subjects and to perform a preliminary assessment of the effect of food on safety and PK parameters of J147. The study will include single ascending dose (SAD) in healthy young and elderly subjects.

Approximately 64 subjects may be included in the study, with an additional 24 to be added depending on the emerging data.

Six cohorts of 8 healthy young male subjects and 2 cohorts of 8 healthy elderly male and female subjects are planned. Depending on emerging safety, tolerability and PK data, 2 additional cohorts of 8 healthy young male subjects in each cohort and 1 additional cohort of 8 elderly male and female subjects may be enrolled.

In each cohort, 6 subjects will be randomized to receive a single dose of J147 orally and 2 subjects will be randomized to receive a matching dose of placebo.

All cohorts will consist of 2 sentinel subjects of whom 1 subject will receive J147 and 1 subject will receive matching placebo. The remaining 6 subjects of whom 5 subjects will receive J147 and 1 subject will receive matching placebo will be dosed at least 24 hours following the sentinel subjects.

Healthy elderly subjects will receive doses that have been found to be safe in healthy young subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntarily agreement to participate in this study and signs an IRB/IEC-approved informed consent prior to performing any of the screening procedures
* Healthy male subjects, between 18 to 50 years of age, inclusive, at the time of signing the informed consent; OR, Healthy male and female subjects, between 60 to 85 years of age, inclusive, at the time of signing the informed consent
* If male, subjects with partners of child bearing potential must be practicing abstinence, part of an abstinent life style or agree to use a highly effective contraception method during the intervention period and for at least 3 months after the last dose of study medication and refrain from donating sperm during this period. Because of the unacceptable failure rate of barrier (chemical and/or physical) methods, the barrier method of contraception must only be used in combination with a highly effective method. Post coital methods of contraception are not permitted.
* If female, must not be pregnant, must not be lactating, and must be of non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or postmenopausal ≥ 1 year.
* Body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive, at screening with a weight of at least 50 kg
* Nonsmokers (or other nicotine use) as determined by history (no nicotine use over the past year) and by urine cotinine concentration (< 200 ng/mL) at the screening visit and admission

Exclusion Criteria:

* Has clinically significant history or evidence of cardiovascular, endocrine, hematologic, immune, gastrointestinal, genitourinary or other body system disease as determined by an Investigator
* Has clinically significant history or evidence of disease or dysfunction in neurological or psychiatric system that is likely to affect the results of the study in the opinion of an Investigator
* Has any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs
* Subject has any concurrent disease or condition that, in the opinion of the Principal Investigator, would make the subject unsuitable for participation in the clinical study
* Has positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV) or human immunodeficiency virus (HIV) antibodies
* Has a urine blood test for ethanol or cotinine at the screening visit or admission
* Has a positive urine drug test (e.g., cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids) at the screening visit or admission
* Females who are breastfeeding
* Is unwilling to or has not avoided consumption of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade or other products containing grapefruit or Seville oranges within 14 days of dosing with study medication
* Has history of alcohol and/or illicit drug abuse within 1 year of entry or is unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to admission until discharge from the clinical unit
* Has donated blood (> 500 mL) or blood products within 30 days prior to first day of dosing
* Requires treatment with any medication, prescription or over-the-counter (OTC) medications (including vitamins [mega doses], dietary supplements or herbal medications), prescription medications within 14 days prior to administration of study medication. By exception, acetaminophen ≤ 1000 mg per day and vitamin products at recommended daily doses are permitted
* Has received any known hepatic or renal clearance altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazines or herbal/plant-derived preparations such as St. John's wort) for a period of 30 days prior to dosing
* Has used an investigational drug within 30 days prior to screening
* Has a history of hypersensitivity or allergies to J147, any components of formulated J147, or any drug within the same class; minor drug allergies to a drug in another drug class may be approved by an Investigator if not considered of clinical relevance
* Has clinically significant abnormal vital signs, 12-lead ECGs, physical examination, clinical laboratory, or other safety variable, as judged by an Investigator
* Is considering or has scheduled any surgical procedure during study participation
* Requires a special diet or has a significant food allergy or intolerance; if the subject or patient is vegetarian, he or she may be enrolled at an Investigator's discretion
* Is unable to understand the protocol requirements, instructions and study related restrictions, the nature, scope and possible consequences of the clinical study
* Is unlikely to comply with the protocol requirements, instructions and study related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study
* Has previously been enrolled in this clinical study or is currently enrolled in another clinical study
* For the elderly subjects, there must be no evidence of cognitive decline that has been greater than expected for age and no evidence of changes in their level of independence in everyday life.
* Is judged by an Investigator or Sponsor to be inappropriate for the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | from pre-dose to 7+/-2 days post dose
  Nature, frequency and severity of adverse events
Number of subjects with abnormal electrocardiogram | from pre-dose to 7+/-2 days post dose
  12-lead electrocardiogram measurement
Incidence of clinically significant changes in serum biomarker levels in a standard serum chemistry panel | from pre-dose to 7+/-2 days post dose
  Changes in standard serum chemistry measures will be assessed.
Incidence of clinically significant changes in hematological biomarker levels in a standard hematology panel | from pre-dose to 7+/-2 days post dose
  Changes in standard hematology measures will be assessed.
Incidence of clinically significant changes in urine biomarker levels in a standard urinalysis panel | from pre-dose to 7+/-2 days post dose
  Changes in standard urinalysis measures will be assessed.
Number of patients exhibiting changes in standard Physical Examination results | from pre-dose to 7+/-2 days post dose
Number of patients exhibiting changes in standard Neurological Examination results | from pre-dose to 7+/-2 days post dose

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 0-48 hours post dose
Time to Cmax (Tmax) | 0-48 hours post dose
Area under the plasma concentration vs. time curve (AUC) | 0-48 hours post dose
Terminal rate constant | 0-48 hours post dose
Terminal half-life (t1/2) | 0-48 hours post dose
Apparent plasma clearance (CL/F) | 0-48 hours post dose
Renal clearance (CLr) | 0-48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kankam, MD, PhD, MPH, Principal Investigator — Vince & Associates Clinical Research, Inc.
Locations (1):
- Vince & Associates Clinical Research, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen Q, Prior M, Dargusch R, Roberts A, Riek R, Eichmann C, Chiruta C, Akaishi T, Abe K, Maher P, Schubert D. A novel neurotrophic drug for cognitive enhancement and Alzheimer's disease. PLoS One. 2011;6(12):e27865. doi: 10.1371/journal.pone.0027865. Epub 2011 Dec 14. PMID 22194796
- [Background] Prior M, Dargusch R, Ehren JL, Chiruta C, Schubert D. The neurotrophic compound J147 reverses cognitive impairment in aged Alzheimer's disease mice. Alzheimers Res Ther. 2013 May 14;5(3):25. doi: 10.1186/alzrt179. eCollection 2013. PMID 23673233
- [Background] Currais A, Goldberg J, Farrokhi C, Chang M, Prior M, Dargusch R, Daugherty D, Armando A, Quehenberger O, Maher P, Schubert D. A comprehensive multiomics approach toward understanding the relationship between aging and dementia. Aging (Albany NY). 2015 Nov;7(11):937-55. doi: 10.18632/aging.100838. PMID 26564964
- [Background] Prior M, Goldberg J, Chiruta C, Farrokhi C, Kopynets M, Roberts AJ, Schubert D. Selecting for neurogenic potential as an alternative for Alzheimer's disease drug discovery. Alzheimers Dement. 2016 Jun;12(6):678-86. doi: 10.1016/j.jalz.2016.03.016. Epub 2016 May 2. PMID 27149904
- [Background] Goldberg J, Currais A, Prior M, Fischer W, Chiruta C, Ratliff E, Daugherty D, Dargusch R, Finley K, Esparza-Molto PB, Cuezva JM, Maher P, Petrascheck M, Schubert D. The mitochondrial ATP synthase is a shared drug target for aging and dementia. Aging Cell. 2018 Apr;17(2):e12715. doi: 10.1111/acel.12715. Epub 2018 Jan 7. PMID 29316249